CLINICAL TRIAL: NCT06323694
Title: Quality of Life, Expectations, Thoughts and Fears of Patients on the Waiting List for Spinal Surgery: a Qualitative Study
Brief Title: Quality of Life, Expectations, Thoughts and Fears of Patients on the Waiting List for Spinal Surgery
Acronym: chirurgia-1
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: University of Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: Attesa chirurgia-1
Record Dates: First submitted 2022-11-10; First posted 2024-03-21 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Spinal Surgery
Keywords: spinal fusion; vertebroplasty; quality of life
MeSH Terms: interventions — Quality of Life

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with vertebroplasty: measuring the quality of life in patients on the waiting list for spinal surgery
  Interventions: Behavioral: quality of life
- Patients with spinal fusion: measuring the quality of life in patients on the waiting list for spinal surgery
  Interventions: Behavioral: quality of life

INTERVENTIONS:
Behavioral: quality of life — data collection through questionnaire and interview

SUMMARY:
The objective of this qualitative prospective observational study is to analyze the cognitive aspect, the emotional-behavioral state and the quality of life of patients during their stay on the waiting list for two categories of lumbar spinal surgery: arthrodesis and percutaneous vertebroplasty.

Hypothesis:

Considering the existing evidence that associates some peculiar psychological components (expectations, beliefs, fears, coping strategies) of the patient and the outcome of spinal surgery, as well as the importance that the waiting time for the intervention assumes for recovery post-operative, this study aims to investigate the subjective perception of one's condition and the waiting period prior to the expected spinal surgery.

This is a qualitative prospective observational study, monocentric with variable sample up to the level of saturation. The blind members are the staff who will listen to the recordings of the interviews and prepare the summary table of the same and the statistical researcher who will perform the analyzes.

The selection of the participants will be carried out in such a way as to ensure a heterogeneous sample in terms of age, sex and experience and as representative as possible of the population studied.

The number of participants in qualitative studies is usually determined by intentional sampling, based on the need to understand the full range of possible responses, to obtain the so-called data saturation.

All patients on the waiting lists of the Department of Spinal Surgery, for vertebral arthrodesis or percutaneous vertebroplasty are considered eligible.

The two types of surgery differ both in the surgical procedure and in the duration of the wait before surgery, which is 1-2 months for vertebroplasty and more than one year for spinal arthrodeses which are not of urgency or priority.

DETAILED DESCRIPTION:
Expectations and personal experiences of the patient regarding the state of illness and the path of treatment undertaken are essential for the overall taking into account of the person. In patients undergoing spinal surgery, it has been shown that these factors can influence both perceived patient satisfaction and post-operative outcomes.

In particular, the catastrophization of pain even before surgery has been shown to predict functional disability, postoperative pain and its chronicity.

The literature also highlights that the time spent on the waiting list by patients elected for spinal surgery can influence postoperative pain outcomes and persistence.

It should also be emphasized that, in comparison with candidates for surgery for other districts (hip, knee), patients hospitalized for spinal surgery arrived at the intervention with worse scores on all scales, both physical and mental.

Numerous qualitative studies have investigated various aspects of the patient's subjective experience after surgery: from the experience related to pre- and post-operative rehabilitation programs, to the perspectives on '' introduction of a healthy lifestyle with physical activity ; from the perception of preparation for surgery, to the experience of Enhanced Recovery After Surgery - ERAS.

Some authors have investigated the experience of the entire care path through qualitative studies, interviewing patients also about preoperative experiences , but always in interviews carried out after the operation.

On the other hand, studies carried out on patients on the waiting list are very rare, focusing on expectations and predictors of outcome.

To date, however, no qualitative studies have directly involved patients on the waiting list to investigate their subjective perception of the quality of life, expectations, emotional state, fears. In particular for two categories of lumbar spinal surgery: arthrodesis and percutaneous vertebroplasty.

The objective of this qualitative prospective observational study is to analyze the cognitive aspect, the emotional-behavioral state and the quality of life of patients during their stay on the waiting list for two categories of lumbar spinal surgery: arthrodesis and percutaneous vertebroplasty.

Hypothesis:

Considering the existing evidence that associates some peculiar psychological components (expectations, beliefs, fears, coping strategies) of the patient and the outcome of spinal surgery, as well as the importance that the waiting time for the intervention assumes for recovery post-operative, this study aims to investigate the subjective perception of one's condition and the waiting period prior to the expected spinal surgery.

This is a qualitative prospective observational study, monocentric with variable sample up to the level of saturation. The blind members are the staff who will listen to the recordings of the interviews and prepare the summary table of the same and the statistical researcher who will perform the analyzes.

The selection of the participants will be carried out in such a way as to ensure a heterogeneous sample in terms of age, sex and experience and as representative as possible of the population studied.

The number of participants in qualitative studies is usually determined by intentional sampling, based on the need to understand the full range of possible responses, to obtain the so-called data saturation.

All patients on the waiting lists of the Department of Spinal Surgery, for vertebral arthrodesis or percutaneous vertebroplasty are considered eligible.

The two types of surgery differ both in the surgical procedure and in the duration of the wait before surgery, which is 1-2 months for vertebroplasty and more than one year for spinal arthrodeses which are not of urgency or priority.

The type of study (qualitative study) is the most suitable for investigating the subjective perception of a problem and its characteristics from a psychosocial point of view.

The semi-structured interview is the most appropriate tool to allow the exploration of the patient's subjective point of view.

The tools to describe patients with respect to catastrophization, convictions with respect to movement, kinesiophobia, anxiety and depression were chosen among the evaluation scales and questionnaires validated in Italian most used in the clinical setting and suggested by consensus of experts In order to facilitate the recruitment process, the selection of subjects will take place in two ways:

1. The patient eligible for the study based on the inclusion and exclusion criteria will be informed about the study by the doctor during the outpatient visit and the insertion who visits him and puts him on the waiting list for the intervention; the investigator will explain to the patient the purpose of the study and will provide him with the form for informed consent.

   Only subjects who have provided their consent will be included in the study.
2. To ensure the recruitment of subjects already included in the list, the staff involved in the study will identify from the waiting list the subjects who meet the inclusion criteria and will recruit them.

These subjects will be contacted by telephone by the researchers of the study 1 month after being placed on the waiting list for vertebroplasty operations and at least 12 months after being placed on the waiting list for arthrodesis operations to organize an individual interview.

The interviews will take place on a date and time established according to individual preferences, to be held at the Rizzoli Orthopedic Institute in a closed room and with no other people present, in addition to the interviewer and the patient.

Before the interview, an initial "booklet" will be delivered, which constitutes the data collection form of the study, including:

* personal and anthropometric data, educational qualifications, work activity and data regarding pain (location and duration);
* the Italian version of the 0-100 Numerical Rating Scale (NRS);
* the Italian version of the Pain Self-Efficacy Questionnaire (PSEQ);
* the Italian version of the Tampa Scale for Kinesiophobia (TSK);
* the Italian version of the Pain Catastrophizing Scale (PCS);
* the Italian version of the Hospital Anxiety and Depression Scale (HADS);
* the Italian version of the Euro Quality of Life Questionnaire (EuroQOL). Once completed, the questionnaires will be placed in a sealed envelope and delivered to the researcher interviewer.

The researcher will carry out the semi-structured interview, without being aware of the results collected during the initial evaluation. The individual interview will aim to investigate the patient's perception of his state of health and quality of life, his beliefs about the surgery, waiting time and recovery, the emotional state related to the pathology and to the intervention.

The in-depth interview will be structured with open questions in order to investigate patients' ideas during the waiting period for surgery, in particular: perceived health and quality of life, emotional state, symptom trend and preparation for intervention, expectations regarding the post-operative period and recovery, fears relating to the intervention and the post-operative phase, fears related to the current health emergency situation.

In order to allow the research promoters to discuss and analyze all the answers to the open questions, the interviews will be audio-recorded with a digital audio recorder and later transcribed anonymously. The interviews will be simultaneously and independently analyzed by at least two members of the study group, in order to reach a consensus on emerging codes and themes. These will be grouped, interpreted and analyzed according to the content analysis method.

Thanks to the emerging design in qualitative research, the analysis will be carried out throughout the period of data collection. Sampling will stop when saturation is reached. The qualitative analysis will then begin with the reading of the transcripts and, based on these transcripts, the analysis of the thematic content will lead to the identification of categories and themes. The data will be analyzed in an iterative way, to refine the evolving themes.

This process will continue until further observations provide new information, thus modifying the categories and themes. These categories will serve as the basis for a final grid, which will then be used to analyze the transcripts. The sample of participants investigated should allow to reach a point where no new categories emerge from the analysis of the transcripts.

Using patient data (generated through interviews) and verification of interpretation by the multidisciplinary team of researchers, the reliability of the data can be verified. This research method is derived from previous similar projects. In the design phase of this study, the researchers and consultants studied the specific topic of the research, in order to reach a better understanding of what will emerge from the participants.

DATA COLLECTION The data necessary for the research will be collected through the questionnaires provided to patients and the interview carried out by the researchers. A special collection report form (CRF) will be used to collect the questionnaire data for each patient enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients on the waiting list for first vertebral arthrodesis or vertebroplasty surgery percutaneous;
* Age over 18;
* Good understanding of spoken and written Italian;
* Obtaining Informed Consent;
* Possibility to go to the Rizzoli Orthopedic Institute on a date to be agreed for carry out the interview with the researchers.

Exclusion Criteria:

* Previous spinal surgery;
* Poor understanding of spoken and written Italian
* Central or peripheral neurological diseases;
* Systemic pathologies;
* Rheumatic pathologies;
* Neuromuscular pathologies;
* Tumors;
* Neuropsychological deficits that do not allow you to fill in the questionnaires and / or answer fully to the interview.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients on the waiting lists of the Dipartiment of Spinal Surgery, for vertebral arthrodesis or percutaneous vertebroplasty are considered eligible.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
Descriptive survey for vertebroplasty patients | after 1 month
  questionnaire on the personal situation of the patient on the waiting list for vertebroplasty
Descriptive survey for spinal arthrodeses patients | after 1 year
  questionnaire on the personal situation of the patient on the waiting list for spinal arthrodeses

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pillastrini P, Ferrari S, Albano A, Beni M, Burbello I, De Cristofaro L, Griffoni C, Mattarozzi K, Nervuti G, Vanti C. Patients' experience on waiting for spinal arthrodesis: a qualitative study. Qual Life Res. 2025 Mar;34(3):833-842. doi: 10.1007/s11136-024-03861-3. Epub 2024 Dec 8. PMID 39648235